CLINICAL TRIAL: NCT04312828
Title: Assessment of Orthopedic Care of the Z-shaped Foot in Children From 6 Months to 2 Years Old
Brief Title: Assessment of Orthopedic Care of the Z-shaped Foot in Infant
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02916-51
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Foot Deformities
MeSH Terms: conditions — Foot Deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orthopedic management of the Z-foot — Orthopedic treatment with femoropedic plasters and slotted splints in 1st intention

SUMMARY:
Real-life, observational, monocentric, ambispective study, carried out in France. The aim of the study is to evaluate the success rate of orthopedic management of the Z-foot after at least 9 months of follow-up.

DETAILED DESCRIPTION:
The study will include a single prospective data collection, which will make it possible to obtain prospective clinical data at the longest follow-up after treatment, with a minimum follow-up of 9 months. This collection will be done during a visit to the office or a phone call, depending on the preference of patients and their parents.

Early data (before the intervention, immediately after, and at 3 months of follow-up) will be collected retrospectively in medical records.

ELIGIBILITY:
Inclusion Criteria:

* Child having presented a congenital idiopathic malformation uni- or bilateral of foot in Z, defined by the presence of an angular adduction of the mid-forefoot and a dorsolateral hump;
* Orthopedic treatment with femoropedic plasters and slotted splints in 1st intention, having started at least 9 months before inclusion;
* Child aged 6 months to 2 years at the start of care;
* Authorization of the parents or the legal representative of the child to collect personal information about their child.

Exclusion Criteria:

* Child having presented a secondary Z foot;
* History of foot surgery;
* Lack of retrospective data to assess the convexity of the external edge of the foot before orthopedic care;
* Inability of the parents or the child's legal representative to understand the study protocol.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who suffered from a congenital idiopathic Z-foot deformation, aged 6 months to 2 years at the time of orthopedic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
The main criterion of the study is the success rate of orthopedic management of the Z-foot. | 9 months
  Success is a composite criterion, measured at the last follow-up, defined by:
  * Outer edge of the straight foot; AND
  * Absence of dorsolateral hump OR possibility of putting on shoes without difficulty AND
  * Absence of recurrence of the malformation OR resumption of surgery OR resumption of orthopedic treatment.

SECONDARY OUTCOMES:
Moderate success rate of the procedure | 9 months
  Defined by an external edge of the foot that is not rectilinear but the possibility of normal footwear, at the greatest distance (relative to the number of feet treated)
Partial and total success rate (relative to the number of patients treated) | 9 months
  * Total success rate: (number of patients with unilateral involvement and foot treated successfully + number of patients with bilateral involvement and both feet treated successfully) / total number of patients.
  * Partial success rate in patients with bilateral involvement: number of patients with only one of the 2 feet treated successfully / number of patients with bilateral involvement.
Convex angle of the outer edge of the foot during follow-up | 9 months
  The evolution of the convexity angle of the external edge of the foot will be studied during treatment and follow-up, in a mixed model with repeated measurements, with the initial severity of the malformation as a cofactor (angle ≤ 15 ° /> 15 ° ).

CONTACTS AND LOCATIONS:
Overall Officials: Mira MD RAMANOUDJAME, Principal Investigator — Clinique Marcel SEMBAT
Locations (1):
- Clinique Marcel SEMBAT, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No